CLINICAL TRIAL: NCT06203600
Title: Randomized Phase II/III Trial of 2nd Line Nivolumab + Paclitaxel + Ramucirumab Versus Paclitaxel + Ramucirumab in Patients With PD-L1 CPS >/= 1 Advanced Gastric and Esophageal Adenocarcinoma (PARAMUNE)
Brief Title: Adding Nivolumab to Usual Treatment for People With Advanced Stomach or Esophageal Cancer, PARAMUNE Trial
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-11064; NCI-2023-11064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2303 (Other: SWOG); S2303 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2024-01-10; First posted 2024-01-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Esophageal Adenocarcinoma; Advanced Gastric Adenocarcinoma; Advanced Gastroesophageal Junction Adenocarcinoma; Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Metastatic Esophageal Adenocarcinoma; Metastatic Gastric Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Unresectable Esophageal Adenocarcinoma; Unresectable Gastric Adenocarcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Nivolumab; Paclitaxel; Taxes; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (nivolumab, ramucirumab, paclitaxel) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 of each cycle, ramucirumab IV over 30-60 minutes on days 1 and 15 of each cycle, and paclitaxel IV over 60 minutes on days 1, 8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and MRI throughout the study. Patients may also optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Drug: Paclitaxel; Other: Questionnaire Administration; Biological: Ramucirumab
- Arm 2 (ramucirumab, paclitaxel) (Active Comparator): Patients receive ramucirumab IV over 30-60 minutes on days 1 and 15 of each cycle and paclitaxel IV over 60 minutes on days 1, 8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and MRI throughout the study. Patients may also optionally undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Other: Questionnaire Administration; Biological: Ramucirumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo optional blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm 1 (nivolumab, ramucirumab, paclitaxel)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Questionnaire Administration — Ancillary studies
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC 1121B; IMC-1121B; IMC1121B; LY 3009806; LY-3009806; LY3009806; Monoclonal Antibody HGS-ETR2

SUMMARY:
This phase II/III trial compares the addition of nivolumab to the usual treatment of paclitaxel and ramucirumab to paclitaxel and ramucirumab alone in treating patients with gastric or esophageal adenocarcinoma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ramucirumab is a monoclonal antibody that may prevent the growth of new blood vessels that tumors need to grow. Paclitaxel is in a class of medications called antimicrotubule agents. It stops cancer cells from growing and dividing and may kill them. Adding nivolumab to ramucirumab and paclitaxel may work better to treat patients with advanced stomach or esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether progression-free survival (PFS) is sufficiently improved in participants randomized to nivolumab + paclitaxel + ramucirumab compared to those randomized to paclitaxel + ramucirumab to warrant a phase III study with overall survival (OS) as the primary endpoint. (Phase II) II. To compare OS in participants randomized to nivolumab + paclitaxel + ramucirumab versus those randomized to paclitaxel + ramucirumab. (Phase III)

SECONDARY OBJECTIVES:

I. To compare PFS between those randomized to nivolumab + paclitaxel + ramucirumab versus those randomized to paclitaxel + ramucirumab. (Phase III) II. To compare OS between participants randomized to nivolumab + paclitaxel + ramucirumab compared to those randomized to paclitaxel + ramucirumab in the event that the trial is completed before the phase III portion.

III. To compare the overall response rate (ORR, including confirmed and unconfirmed, complete, and partial response, according to Response Evaluation Criteria in Solid Tumors [RECIST 1.1] criteria) between those randomized to nivolumab + paclitaxel + ramucirumab compared to those randomized to paclitaxel + ramucirumab among participants with measurable disease.

IV. To compare the overall disease control rate (DCR = ORR + stable disease) between those randomized to nivolumab + paclitaxel + ramucirumab compared to those randomized to paclitaxel + ramucirumab among participants with measurable disease.

V. To evaluate the safety and tolerability of each treatment regimen. VI. To compare health-related quality of life (QOL) by treatment arm at 8 weeks after randomization, measured using the Functional Assessment of Cancer Therapy - Gastric (FACT-Ga) Trial Outcome Index (TOI).

VII. To compare health-related QOL between treatment arms at 8 weeks after randomization using the FACT-Ga total score.

VIII. To compare longitudinal changes in health-related QOL between treatment arms using FACT-Ga TOI up to 24 weeks after randomization.

IX. To compare patient-reported symptoms using selected Patient-Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) items including gastrointestinal as well as constitutional symptoms of fatigue, anorexia, and weight loss between treatment arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle, ramucirumab IV over 30-60 minutes on days 1 and 15 of each cycle, and paclitaxel IV over 60 minutes on days 1, 8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan and magnetic resonance imaging (MRI) throughout the study. Patients may also optionally undergo blood sample collection on study.

ARM 2: Patients receive ramucirumab IV over 30-60 minutes on days 1 and 15 of each cycle and paclitaxel IV over 60 minutes on days 1, 8 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and MRI throughout the study. Patients may also optionally undergo blood sample collection on study.

After completion of study treatment, patients are followed up at 30, 60, 90 days and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have advanced or locally unresectable gastric, gastroesophageal junction or esophageal adenocarcinoma
* Participants must have PD-L1 CPS (Combined Positive Score) ≥ 1. This test would have been performed as part of standard of care (SOC) pathology testing, using tissue obtained within two years prior to registration and collected prior to or after a frontline regimen
* Participants must have a histologically confirmed diagnosis of microsatellite stable (MSS) and HER2 negative gastric, gastroesophageal junction, or esophageal adenocarcinoma
* Participants must have documented unresectable and/or metastatic disease on CT or MRI imaging completed prior to registration. Imaging must have been completed within 28 days prior to registration for participants with measurable disease. CT scans or MRIs used to assess non-measurable disease must have been completed within 42 days prior to registration. All disease must be assessed and documented on the Baseline Tumor Assessment Form
* Participants with treated brain metastases must have no evidence of progression on the follow-up brain imaging after central nervous system (CNS)-directed therapy. All treatment for brain metastases must have been completed at least 28 days prior to registration
* Participants must have disease progression or intolerance to frontline standard of care (SOC) chemotherapy plus either nivolumab, pembrolizumab or any other PD-1 or PD-L1 inhibitor. Peri-operative chemotherapy plus nivolumab, pembrolizumab or any other PD-1 or PD-L1 inhibitor will count as one line if disease progression occurs while on the therapy or within 6 months of completing the chemotherapy plus nivolumab or pembrolizumab or other PD-1/PD-L1 inhibitor cycle
* Participants must not have received more than one prior line of systemic therapy defined as chemotherapy plus either nivolumab, pembrolizumab, or any other PD-1 or PD-L1 inhibitor, in the stage IV or unresectable setting. Peri-operative or adjuvant nivoluamb or other PD-1/PD-L1 inhibitors would count as one prior line of systemic therapy if patients progressed while on nivolumab (or other PD-1/PD-L1 inhibitors) or within 6 months of stopping it

  * Note: Radiation or any other regional therapy options done to address local residual disease or metastatic disease would not count as a line of therapy. Maintenance therapy with a different form of fluoropyrimidine (i.e. switching from capecitabine to fluorouracil [5FU]) would not count as another line of therapy
* Participants must not have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Participants are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if < 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted, as long as there has been a washout period for corticosteroids of ≥ 7 days prior to registration
* Participants must not have prior significant immunotherapy related adverse events requiring permanent discontinuation of the immunotherapy agent including events like pneumonitis, myocarditis, renal failure, Guillain barre syndrome, or myasthenia gravis. Participants with endocrinopathy events leading or not to replacement steroids, thyroid hormone, insulin, or cortisol are eligible
* Participants must not have received a live attenuated vaccination within 28 days prior to registration
* Participants must not have had a major surgery within 28 days or subcutaneous venous access device placement within 7 days prior registration
* Participants must have fully recovered from the effects of prior surgery in the opinion of the treating investigator. Any participants with postoperative bleeding complications or wound complications from a surgical procedure performed in the last eight weeks should be excluded
* Participants must not have plans to undergo elective or planned major surgery during the clinical trial
* Participants must not have active bleeding or prior history of gastrointestinal (GI) perforation, fistula or significant GI bleeding (requiring transfusion, endoscopic or surgical intervention) within 84 days prior to registration
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, investigational agents, biologic or hormonal therapy for cancer treatment while receiving treatment on this study
* Participants must not have a history of a grade 3 or 4 allergic reaction attributed to humanized or human monoclonal antibody therapy
* Participants must not have a history of grade 3 or 4 immunotherapy related toxicities with the exception of hormonal abnormalities like thyroiditis or thyroid derangements
* Participants must be ≥ 18 years old
* Participants must have Zubrod Performance Status of 0-2
* Participants must have a complete medical history and physical exam within 28 days prior to registration
* Leukocytes ≥ 2 x 10^3/uL (within 28 days prior to registration)
* Absolute neutrophil count ≥ 1.2 x 10^3/uL (within 28 days prior to registration)
* Hemoglobin ≥ 9.0 g/dL (within 28 days prior to registration)
* Platelets ≥ 100 x 10^3/uL (within 28 days prior to registration)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to registration) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 × institutional ULN (within 28 days prior to registration) (unless liver metastases are present, in which case they must be ≤ 5 x ULN)
* Participants must have a calculated creatinine clearance ≥ 40 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration
* Participants' urinary protein must be ≤ 1+ on dipstick or routine urinalysis (UA) within 28 days of registration. Random analysis of urine protein with a normal value is sufficient. If urine dipstick or routine analysis indicated proteinuria ≥ 2+, then a 24-hour urine is to be collected and demonstrate < 1000 mg of protein in 24 hours to allow participation in the study
* Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2 or better
* Participants must have recovered to baseline or < grade 2 CTCAE version (v) 5.0 from toxicities related to any prior treatments, unless AE(s) are clinically stable on supportive therapy
* Participants must not have experienced arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to registration
* Participants must not have uncontrolled blood pressure within 28 days prior to registration as determined by the treating investigator
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load on the most recent test results obtained within 6 months prior to registration
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must not have a history of inflammatory bowel disease, (including ulcerative colitis and Crohn's disease), symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and myasthenia gravis, multiple sclerosis). Note: Participants with Graves' disease will be allowed
* Participants must not have a history of pneumonitis that has required oral or IV steroids within the last 12 months prior to registration
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants who can complete patient reported outcomes (FACT-Ga and PRO-CTCAE) questionnaires in English or Spanish must participate in the quality of life studies
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Phase II) | From date of randomization to date of first documentation of progression or symptomatic deterioration or death due to any cause, assessed up to 3 years
  The distribution of PFS will be estimated using the method of Kaplan-Meier and compared using a 1-sided stratified log-rank test.
Overall survival (OS) (Phase III) | From date of randomization to date of death due to any cause, assessed up to 3 years
  The distribution of OS will be estimated using the method of Kaplan-Meier and compared using a 1-sided stratified log-rank test.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  Will be compared across arms in participants with measurable disease via Fisher's exact test.
Disease control rate (DCR) | Up to 3 years
  DCR = ORR + stable disease per Response Evaluation Criteria in Solid Tumors 1.1. Will be compared across arms in participants with measurable disease via Fisher's exact test.
Incidence of adverse events | Up to 3 years

OTHER OUTCOMES:
Disease-free survival (DFS) | Up to 3 years
  The hazard ratio of DFS and the corresponding 95% confidence intervals will be estimated for subgroups defined by sex, race, and ethnicity, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Anwaar Saeed, Principal Investigator — SWOG Cancer Research Network
Locations (366):
- United States (366):
  - Baptist Health Medical Center - Little Rock, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - AdventHealth Orlando, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Mercyhealth Cancer Institute - Rockford, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - UPMC Western Maryland, Cumberland, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Cone Health Cancer Center at Asheboro, Asheboro, North Carolina
  - Cone Health MedCenter Asheboro, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Saeed A, Colby S, Oberstein PE, Duda DG, Park R, Agarwal R, Figueroa-Moseley C, Vaidya R, Unger JM, Guthrie KA, Rocha FG, Senthil M, Safyan RA, Wainberg ZA, Iqbal S, Chiorean EG, Philip PA. S2303: phase II/III trial of paclitaxel + ramucirumab +/- nivolumab in gastric and esophageal adenocarcinoma (PARAMUNE). Future Oncol. 2025 May;21(11):1325-1331. doi: 10.1080/14796694.2025.2485020. Epub 2025 Mar 28. PMID 40155326